CLINICAL TRIAL: NCT05769595
Title: A Single-dose Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-2060 in Japanese Older Participants With End-stage Renal Disease on Dialysis.
Brief Title: Single Dose Study of MK-2060 to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Older Japanese Participants on Dialysis (MK-2060-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2060-012; MK-2060-012 (Other: Merck); jRCT2041230025 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: End-Stage Renal Disease (ESRD); End-Stage Kidney Disease (ESKD); Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MK-2060 (Experimental): Participants receive MK-2060 50 mg via a single intravenous (IV) infusion over 60-minutes.
  Interventions: Biological: MK-2060
- Placebo (Placebo Comparator): Participants receive a single IV saline infusion over 60 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: MK-2060 — Lyophilized powder diluted in normal saline for IV infusion
  Arms: MK-2060
Drug: Placebo — IV infusion
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of MK-2060 after a single dose intravenous (IV) administration in Japanese older participants with end stage renal disease (ESRD) on dialysis. There is no primary hypothesis for this study.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Japanese descent with all 2 biological parents of Japanese descent
* On hemodialysis (HD) or hemodiafiltration (HDF) with single-pool Kt/V (spKt/V) ≥1.2, using arteriovenous (AV) fistula or AV graft ≥3 months prior to Screening 1 at a healthcare center, and is on the same dialysis regimen ≥2 weeks prior to Screening 1
* Be judged to plan to continue or anticipate the use of the current AV fistula or AV graft until the poststudy visit

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* On peritoneal dialysis or other dialysis modalities except for HD and HDF
* History of deep vein thrombosis or pulmonary embolism
* History of vascular access thrombosis within 1 month prior to Screening 1
* Personal or family history of bleeding disorder
* History of GI bleeding, duodenal polyps or active gastroduodenal ulcer within 5 years prior to Screening 1, or history of severe hemorrhoidal bleed within 3 months prior to Screening 1
* History of frequent epistaxis within 3 months prior to Screening 1 or active gingivitis
* At the time of screening or predose, planned significant dental procedures, or other planned surgical procedures within duration of participation in the trial
* History of receiving any human immunoglobulin preparation such as intravenous immunoglobulin (IVIG) or a brand of Rho(D) immune globulin (RhoGAM) within 1 year prior to Screening 1
* History of receiving any biological therapy within 3 months prior to Screening 1, or vaccination within 1 month prior to the dose of study intervention
* Requires or anticipates requiring the use of following prohibited medications until the poststudy visit: anticoagulants, antiplatelet medications and non-steroidal anti-inflammatory drugs (NSAIDs)
* Participated in another investigational study within 1 month prior to Screening 1
* Has blood coagulation test (activated partial thromboplastin time [aPTT] or prothrombin time [PT]) above 1.2X upper limit of normal (ULN) at Screening 1 from the central laboratory for safety

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (12):
- Japan (12):
  - Kasugai Municipal Hospital ( Site 1203), Kasugai, Aichi-ken
  - Chubu Rosai Hospital ( Site 1202), Nagoya, Aichi-ken
  - Kojunkai Daido Hospital ( Site 1207), Nagoya, Aichi-ken
  - Jomo Ohashi Clinic ( Site 1210), Maebashi, Gunma
  - Ibaraki Prefectural Central Hospital ( Site 1211), Kasama, Ibaraki
  - Shonan Kamakura General Hospital ( Site 1205), Kamakura, Kanagawa
  - Matsumoto City Hospital ( Site 1209), Matsumoto, Nagano
  - Keiaikai Nakamura Hospital ( Site 1213), Beppu, Oita Prefecture
  - Omi Fureai Hospital ( Site 1204), Kusatsu, Shiga
  - Ikegami General Hospital ( Site 1206), Ōta-ku, Tokyo
  - Japanese Red Cross Fukuoka Hospital ( Site 1214), Fukuoka
  - Yamagata Tokushukai Hospital ( Site 1201), Yamagata

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-2060: Participants received MK-2060 50 mg via a single intravenous (IV) infusion over 60 minutes.
- Placebo: Participants received a single IV saline infusion over 60 minutes.
Period: Overall Study
Arm/Group | MK-2060 | Placebo
Started | 12 | 5
Completed | 12 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-2060 | Placebo | Total
Number analyzed (Participants) | 12 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (7.2) | 66.2 (8.3) | 69.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 5 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 5 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who experienced an AE is reported.
Time Frame: Up to approximately 164 days
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- MK-2060: Participants received MK-2060 50 mg via a single IV infusion over 60 minutes.
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 5
Participants | 10 | 4

2. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who discontinued study due to an AE is reported.
Time Frame: Up to approximately 164 days
Population: All participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 5
Participants | 0 | 0

3. Secondary Outcome: Area Under the Concentration-Time Curve of MK-2060 From Time 0 to Infinity (AUC 0-inf)
Description: Blood samples were collected at specified intervals for the determination of AUC0-inf. AUC0-inf is defined as the area under the concentration-time curve of MK-2060 from time zero to infinity.
Time Frame: Predose, 1, 12, 24, 48 and 52 hours postdose; 5, 12, 15, 22, 60, 90, and up to 157 days post dose; and twice daily on Days 8, 29, 120: pre- and post-dialysis
Population: All participants who were compliant with the study procedures and have available data from at least one MK-2060 treatment were included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nmol/L
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
hours*nmol/L | 35000 (31.8) |

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve of MK-2060 From Time 0 to Last (AUC0-last)
Description: Blood samples were collected at specified intervals for the determination of AUC0-last. AUC0-last is defined as the area under the plasma concentration-time curve from time zero to time of last measurable concentration of MK-2060.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nmol/L
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
hours*nmol/L | 34500 (31.8) |

5. Secondary Outcome: Area Under the Concentration-Time Curve of MK-2060 From Time 0 to 168 Hours Postdose (AUC0-168)
Description: Blood samples were collected at specified intervals for the determination of AUC0-168. AUC0-168 is defined as the area under the concentration-time curve of MK-2060 from time zero to 168 hours.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nmol/L
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
hours*nmol/L | 10100 (23.4) |

6. Secondary Outcome: Maximum Concentration (Cmax) of MK-2060
Description: Blood samples were collected at specified intervals for the determination of Cmax. Cmax is defined as the maximum concentration of MK-2060 reached.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
nmol/L | 110 (26.0) |

7. Secondary Outcome: Concentration at 168 Hours (C168) Postdose of MK-2060
Description: Blood samples were collected at specified intervals for the determination of C168. C168 is defined as the maximum concentration of MK-2060 reached at 168 hours postdose.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- MK-2060: Participants received MK-2060 50 mg via a single intravenous (IV) infusion over 60-minutes.
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
nmol/L | 39.0 (30.9) |

8. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-2060
Description: Blood samples were collected at specified intervals for the determination of Tmax. Tmax is defined as time to the maximum concentration of MK-2060 reached.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
hours | 1.03 [0.88 to 12.02] |

9. Secondary Outcome: Time of the Last Measurable Plasma Concentration (Tlast) of MK-2060
Description: Blood samples were collected at specified intervals for the determination of Tlast. Tlast is defined as the time to the last measurable concentration of MK-2060 reached.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
hours | 3407.34 [2186.65 to 3695.18] |

10. Secondary Outcome: Terminal Half-Life (t ½) of MK-2060
Description: Blood samples were collected at specified intervals for the determination of t½. t½ is defined as the time required to divide the MK-2060 plasma concentration by two after reaching pseudo-equilibrium, following a single dose of MK-2060.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
Days | 22.7 (18.2) |

11. Secondary Outcome: Clearance (CL) of MK-2060
Description: Blood samples were collected at specified intervals for the determination of CL. CL is the volume of plasma from which the study drug is completely removed per unit time.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
Liters/hour | 0.00964 (31.8) |

12. Secondary Outcome: Volume of Distribution (Vz) of MK-2060
Description: Blood samples were collected at specified intervals for the determination of Vz. Vz is the apparent volume of distribution during the terminal phase.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 0
Liters | 7.58 (28.5) |

13. Secondary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (aPTT)
Description: Blood samples were collected for the determination of aPTT. Change from baseline in aPTT up to 168 hours post dose (pre dialysis) is reported.
Time Frame: Baseline and 168 hours post dose
Population: All participants who were compliant with the study procedures and have available data from at least one treatment were included.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold-Change from baseline
Arm/Group | MK-2060 | Placebo
Number analyzed (Participants) | 12 | 5
Fold-Change from baseline | 2.45 [2.27 to 2.63] | 0.97 [0.87 to 1.09]
Statistical Analysis 1: Comparison: MK-2060 vs Placebo; Test type: Other; Geometric Mean Ratio = 2.51, 90% CI 2-sided [2.24 to 2.82] — Geometric mean ratio is MK-2060/placebo

ADVERSE EVENTS:
Time Frame: Up to approximately 164 days
Description: All participants who received at least one dose of treatment.
Groups:
- MK-2060 50 mg: Participants received MK-2060 50 mg via a single intravenous (IV) infusion over 60 minutes.
Arm/Group | MK-2060 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/12 | 1/5
Other Adverse Events (participants affected / at risk) | 9/12 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2060 50 mg (N=12) | Placebo (N=5)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-2060 50 mg (N=12) | Placebo (N=5)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt stenosis (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Bleeding time prolonged (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (2)
Internal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT05769595/Prot_SAP_000.pdf